CLINICAL TRIAL: NCT06644430
Title: Ablation of Pulmonary Oligometastasis Combined With System Compared System Therapy for Advanced Hepatocellular Carcinoma: a Multicenter Retrospective Study
Brief Title: Ablation of Pulmonary Oligometastasis Combined With System for Advanced Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Other Study IDs: CHEST-002
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Advanced Hepatocellular Carcinoma; Lung Cancer; Oligometastasis; Ablation; Systemic Therapy
Keywords: Advanced hepatocellular carcinoma; Lenvatinib; Sorafeinib; Camrelizumab; Tislelizumab; Sintilimab; Toripalimab; Apatinib
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ablation+system group: Participants received ablation of plumonary combined systemic therapy
  Interventions: Procedure: Ablation; Drug: system therapy
- System group: Participants received systemic therapy
  Interventions: Drug: system therapy

INTERVENTIONS:
Procedure: Ablation — Ablation including (microwave ablation, radiofrequency ablation, cryoblation), this surgery was conducted under CT guidence. The pulmonary was completely ablated.
  Groups: Ablation+system group
Drug: system therapy — Paticipants received systemic therapy according the instructions.

SUMMARY:
Ablation has been an effective therapy in treating intrathoracic metastases. However, for hepatocellular carcinoma with pulmonary oligometastasis, ablation of metastases remains relatively unexplored and still needs clinical evidence.

DETAILED DESCRIPTION:
Systemic therapy is the standard treatment for advanced hepatocellular carcinoma (HCC) with metastasis. However, metastases with limited number (oligometastasis) can represent a subtype and transition point between localized disease and widespread metastases. Thus, eliminating metastases could be advantageous and beneficial to the prognosis if feasible and permitted. Image-guided ablation therapy, such as microwave ablation (MWA), radiofrequency ablation (RFA), and cryoablation, has attracted great interest as a minimally invasive approach against intrathoracic metastases. Recently, ablation has been used on patients with pulmonary metastases from various cancers. This technique yields high proportions of sustained complete responses and is associated with relatively low morbidity. This multicenter study focuses on the management of ablation of oligometastasis therapy combined with systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of primary HCC, confirmed histologically or clinically according to the criteria of the American Association for the Study of Liver Diseases;
2. presence of pulmonary oligometastasis, the metastases found within three month of HCC diagnosis;
3. metastases with limited five sites and no more two organs involved, with a maximum diameter of ≤5cm;
4. receipt of first-line systemic therapy for minimum of 3 months before ablation, with controlled intrahepatic tumors and no progression of metastases. Controlled intrahepatic tumors were defined as those showing a partial or stable response according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST);
5. undergone locoregional treatments, including transarterial artery chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC) were included;
6. classified as Child-Pugh class A or B and having an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. no history of other malignancies.
8. life expectancy more than 3 months;
9. agreed to participated in this clinical trial;
10. Hemameba ≥3.0 x109/L, neutrophil ≥1.5x109/L, hemoglobin≥10.0 g/L, platelet≥100x 109/L, ALT; AST; bilirubin ≤1.5-fold normal, GFR≥60ml/min.

Exclusion Criteria:

1. intermediate HCC;
2. age < 18 years or > 75 years;
3. advanced HCC with more than five metastases;
4. no response to Lenvatinib;
5. metastases size > 5 cm;
6. life expectancy less than 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thermal ablation, as a minimal therapy, has been recommended as a favorable therapy for metastases worldwide. However, for advanced hepatocellular carcinoma with pulmonary oligometastasis, the standard of care is system therapy. However, the evidence of ablating the oligometastasis is limited. In this multicenter study, we want to indicate that compared with systemic therapy, patients received thermal ablation of pulmonary oligometastasis plus system therapy showed significantly longer survival. This study will supplement the current situation where system therapy is the standard of care for hepatocellular carcinoma with oligometastasis.
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | 12 months
  Progression was defined as progressive disease by independent radiologic review

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  OS is the length of time from the date of inclusion until death from any cause.
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response is either a complete response or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided